CLINICAL TRIAL: NCT03964376
Title: Nasal High Flow Therapy Versus Postoperative Usual Care in Surgical Patients with Unrecognized Obstructive Sleep Apnea: a Randomized Controlled Trial (A PHASE 2 STUDY)
Brief Title: Nasal High Flow Therapy in Surgical Patients with Unrecognized Obstructive Sleep Apnea
Acronym: POSAII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-5980
Record Dates: First submitted 2019-01-07; First posted 2019-05-28 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea; Sleep Disordered Breathing
Keywords: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nasal High Flow Group (Experimental): Nasal High-Flow oxygen delivery will be applied starting at airflow of minimum 20 Litre/minute. It will be titrated in 15Litre/minute increments to 35 Litre/minute and a maximum 50 Litre/minute as determined by patient comfort. O2 supplementation will be managed by the anesthesia and surgical health care team to maintain the oxygen saturation level in the blood between 92-95%. In the Nasal High-Flow group, when SPO2 is in the range of 92-95%, air will be given instead of oxygen for the 1st 3 nights and during the day, if required, till discharge, whichever is earlier.
  Interventions: Other: Nasal High Flow
- Usual Care Group (Other): In the usual care, patients will receive oxygen at 2-4 Litre/minute via nasal cannula or 6 Litre/minute via facemask titrated to keep SpO2 level in the range of 92-95%. When SpO2 level reaches in the range of 92-95%, oxygen delivery will be discontinued.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Nasal High Flow — Delivery of oxygen via OptiflowTM system (AirvoTM, Fisher & Paykel Inc.) with airflow of 20 to 50 Litre/minute
  Arms: Nasal High Flow Group
Other: Usual Care — Delivery of oxygen at 2-4 Litre/minute via nasal cannula or 6 Litre/minute via face mask
  Arms: Usual Care Group

SUMMARY:
In this study the investigators will determine whether using high flow oxygen in moderate-to-severe Obstructive Sleep Apnea patients following a major non cardiac surgery is more efficacious than usual care in preventing decrease in oxygen level in blood.

DETAILED DESCRIPTION:
The POSA-II trial is a culmination of the investigator's program of research to prevent postoperative adverse outcomes in surgical patients with untreated Obstructive Sleep Apnea (OSA). It is a multi center open label, randomized clinical trial of nasal high-flow vs. usual care in patients with untreated moderate-to-severe OSA undergoing major non cardiac surgery. It is a proof of concept trial to show that nasal high-flow reduces severe desaturation, the causal mechanism for OSA-related adverse events, and to collect key feasibility data for a large international multi center trial with enough power to detect effects on the clinical outcomes. Eligible patients undergoing major non cardiac surgery with high-risk OSA will have a home sleep study. One hundred and ninety patients with moderate-to-severe Sleep Apnea will be randomized into either nasal high-flow or usual care group. Sleep studies, oximetry, electrocardiogram (ECG), and Troponin will be done preoperatively. Postoperatively, ECG and Troponin will be determined daily for the 1st three days, and nocturnal oximetry for the 1st 3 nights. Patients will be followed during their hospitalization and for 30 days postoperatively to ascertain any adverse outcomes. A blinded clinical events committee will adjudicate all components of the composite outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age ≥45 years, undergoing major elective non cardiac surgery under general and/or regional anesthesia with anticipated overnight stay or longer in hospital
* Patients with untreated moderate-to-severe Obstructive Sleep Apnea.
* STOP-Bang score 5 or higher

Exclusion Criteria:

* Predetermined need for postoperative CPAP therapy or ventilation,
* Cheyne-Stokes respiration or Central Apnea,
* Oxygen dependent due to moderate to severe chronic obstructive lung disease available Forced Expiratory Volume at 1 second of < 50% predicted) or advanced interstitial lung disease,
* Pre-existing chronic hypercapnia or obesity hypoventilation syndrome, Intracranial and otolaryngological procedures, and
* Unable to use nasal high-flow (nasal/oral malformations, pre-existing tracheostomy, planned postoperative nasal packing).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Oxygen Desaturation Index (ODI) | 72 hours
  The investigators will measure Oxygen Desaturation Index(the number of desaturation events per hour) by using Pulsox 300i for maximum of three nights post-operatively at the hospital preventing the severe desaturation in surgical patients with untreated moderate-to-severe OSA undergoing major non cardiac surgery. Higher values of ODI are considered worst. If successful, it will provide feasibility data for the performance of a large randomized clinical trial focusing on clinical outcomes and the cost effectiveness of the therapy to the health care system.

SECONDARY OUTCOMES:
Time (minutes) spent below 90% and 80% SpO2 (T90, T80) | 72 hours
  The investigators will measure the time spent in minutes with SpO2 between 0% to %79 (T80) and the time spent in minutes with SpO2 between 0% to 89% (T90). ODI, T90 and T80 will serve as surrogate outcomes of adverse events in the pilot study. In POSA study, an increase in time spent with SpO2 <80% after surgery was associated with a higher risk of postoperative vascular events under usual care.
Compliance to Nasal High-Flow | 72 hours
  To determine the tolerability and adherence of patients with OSA to Nasal High-Flow in the wards using a 10-point numeric rating scale to grade general discomfort, in which points 0 to 3 means not comfortable, 4 to 6 means comfortable and 7 to 10 means the most comfortable.
Titration protocol of nasal high-flow | 72 hours
  The appropriate titration protocol of nasal high-flow will be measured; FiO2: flow rates.
The rate of postoperative adverse events | 30 days
  The rate of postoperative cardiovascular events will be collected during hospitalization and following discharge from hospital, emergency department (if visited) and physician records, and patient by phone at day 30. Adjudicators who are blinded to the results of the ECG, Troponin, sleep study and oximetry will evaluate outcome events.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MBBS FRCPC, Principal Investigator — University of Toronto/ University Health Network
Locations (8):
- Canada (3):
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hopsital, Dept. of Anesthesia, Toronto, Ontario
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Malaysia (2):
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- Singapore (2):
  - Khoo Teck Puat Hospital, Singapore
  - Singapore General Hospital, Singapore